CLINICAL TRIAL: NCT06214247
Title: A Prospective, Open Label, Multi-center, Randomized Study Designed to Evaluate the Safety and Efficacy of Scoring PTCA Catheter on Subjects During Percutaneous Coronary Intervention
Brief Title: Wedge NC - Scoring Balloon Dilatation Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 814
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Wedge NC Scoring Balloon Dilatation Catheter in the test group, subsequently completing the remaining procedure.
  Interventions: Device: Wedge NC Scoring Balloon Dilatation Catheter
- Control Group (Experimental): During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using a similar product(Scoring Balloon Dilatation Catheter) on the market in the control group, subsequently completing the remaining procedure.
  Interventions: Device: Scoreflex Scoring Balloon Dilatation Catheter

INTERVENTIONS:
Device: Wedge NC Scoring Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Wedge NC Scoring Balloon Dilatation Catheter in the test group, subsequently completing the remaining procedure.
  Arms: Test Group
Device: Scoreflex Scoring Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using a similar product on the market in the control group, subsequently completing the remaining procedure.
  Arms: Control Group

SUMMARY:
To evaluate the efficacy and safety of Wedge NC Scoring Balloon Dilatation Catheter for dilating coronary stenosis during PCI in comparison with a similar product on the market.

DETAILED DESCRIPTION:
The prospective, multicenter, open-label, randomized clinical study is designed to verify the efficacy and safety of Wedge NC Scoring Balloon Dilatation Catheter in the application of dilatating coronary artery stenosis during PCI in comparison with a similar product on the market. The study is planned to enroll 198 subjects, who are randomly assigned to the test group (99 cases) and the control group (99 cases).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Subjects must have a single or double vessel coronary artery disease (CAD) and clinical evidence of ischemic heart disease, such as CAD, stable / unstable angina or silent ischemia.
3. Subjects with coronary artery stenosis confirmed by imaging examination are suitable for percutaneous coronary intervention (PCI).
4. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
5. Subject must have de novo or restenotic lesion(s) in native coronary arteries, including in-stent restenosis suitable for percutaneous coronary intervention.
6. Target lesion with reference vessel diameter (RVD) of 2.0mm - 4.0mm, length ≤30mm (by visual inspection).
7. Only one lesion will be selected as the target lesion for revascularization when subjects have multiple lesions requiring treatment. Tandem lesions (defined as multiple lesions) are deemed one lesion if they can be covered by a single stent.
8. If target lesions and non-target lesions are treated simultaneously, they must be located in different coronary artery from the Target lesion

Exclusion Criteria:

1. Subjects with bleeding tendency, contraindications to antiplatelet agent and anticoagulant therapy, and inability to anticoagulant therapy.
2. Subjects are sensitivity to contrast media which cannot be adequately pre-medicated.
3. Subjects with severe renal failure, whether on dialysis or not, with a glomerular filtration rate (eGFR) level < 30ml/min/1.73m2 or serum creatinine level> 2.0 mg/dl within 7 days prior to index procedure.
4. Subjects with decompensated congestive heart failure or cardiogenic shock.
5. Subjects with expected life less than 12 months.
6. Subjects with an active peptic ulcer or active gastrointestinal bleeding within 1 month prior to index procedure.
7. Subjects with an embolic stroke or transient ischemic attack within 2 months prior to index procedure.
8. Subject with known pregnancy or is nursing. Women of child-bearing potential shall undertake a pregnancy test before index procedure.
9. Subjects enrolled in any other clinical trial within 1 month prior to the trial or currently.
10. Subjects who have poor compliance and cannot complete the trial as required.
11. Lesions with total coronary artery occlusion (TIMI 0 or 1).
12. Severe calcifications (grade Ⅲ-Ⅳ) or extreme angulation (>90°), etc., and lesions are inability to pass the study balloon or stent.
13. Lesions with visible thrombosis or ulcers.
14. Lesions with significant intima tears.
15. Unprotected left main disease.
16. Lesions located within an artery/saphenous vein graft or graft anastomosis.
17. Coronary artery spasm without significant stenosis.
18. Saphenous vein graft degenerative disease
19. Other situations that the investigator considers inappropriate for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Procedure Success Rate | before discharge or within 3 days after the procedure
  Procedure success is defined as the target lesion residual stenosis ≤30% right after PCI, without death, Q-wave or non-Q-wave myocardial infarction, or emergency coronary artery bypass grafting (CABG) during postoperative hospitalization.

SECONDARY OUTCOMES:
Clinical Success Rate | 30-day follow-up after procedure
  Clinical success is defined as the composite endpoint of no Major Adverse Cardiovascular Events (MACE) at follow-up, including cardiac death (also considered cardiac death if the cause of death is uncertain), target vessel myocardial infarction (TV-MI) and target lesion revascularization (TLR)
Device Procedural Success Rate | Immediately after procedure
  The following conditions need to be met for the successful balloon dilatation of stenotic lesions:
  1. Successful delivery, inflation, deflation, and withdrawal of the study balloon.
  2. No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in Thrombolysis In Myocardial Infarction (TIMI) flow from baseline as related to the study balloon
Minimum Luminal Diameter (MLD) | Immediately after procedure
  The minimal diameter of the target lesion, evaluated by quantitative coronary analysis (QCA).
Percent of Diameter Stenosis(%DS) | Immediately after procedure
  %DS = (RVD - MLD) / RVD × 100%, MLD refers to the immediately postoperative minimum luminal diameter, RVD refers to the reference vessel diameter.
Acute Lumen Gain (ALG) | Immediately after procedure
  ALG = immediately postoperative MLD - preoperative MLD
Balloon Slippage Rate | Immediately after procedure
  Balloon slippage is defined as a forward or backward movement of the balloon of at least 3mm during its inflation at the lesion site
Surgical complication | Day 0
  Incidence of Complications in a Single Operation
Rate of Adverse Events | Month 3
  Adverse events include death (cardiogenic death or non-cardiogenic death), acute myocardial infarction (Q wave or non-Q wave), target lesion revascularization (TLR), target vessel revascularization (TVR), other cardiac surgery and other cardiac adverse events, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (11):
- China (11):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Dongguan Tongwah Hospital, Dongguan, Guangdong
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hangzhou First People's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Xu J, Chen D, Gao F, Liu Y, Cui H, Wang J, Guo S, Du Z, Huang J, Zhang X, Jiang W, Cheng Z, Jiang J. Randomized study assessing the effectiveness and safety of a novel scoring balloon for percutaneous coronary intervention: the Wedge NC trial. J Thorac Dis. 2025 Apr 30;17(4):2101-2112. doi: 10.21037/jtd-24-1457. Epub 2025 Apr 27. PMID 40400945